CLINICAL TRIAL: NCT00363012
Title: Development of HER-2/Neu (HER2) ICD Memory Immunity After Vaccination With a Plasmid Encoding HER2 ICD in Patients With Advanced Stage HER2 Overexpressing Breast and Ovarian Cancers
Brief Title: Immune Response in Patients Who Have Undergone Vaccine Therapy for Stage III or Stage IV Breast Cancer That Overexpresses HER2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Principal Investigator, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6271; P30CA015704 (NIH); K23CA100691 (NIH); UWCC-6271; UWCC-03-6843-D03; UWCC-117; FHCRC-6271; CDR0000492707 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Flow Cytometry; Immunohistochemistry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: HER-2/neu intracellular domain protein — 300mcg (100mcg/peptide) of the HER2 ICD peptide mixture per skin test. This will be injected intradermally on the back at 6 months post active immunization.
Other: flow cytometry — This is a laboratory test used to assess the antigen specific T cell population.
Other: immunohistochemistry staining method — This is a laboratory test used to identify CD3+, CD4+, CD45R0+, CD8+, and DC1a+ present in the skin biopsy.
Procedure: biopsy — A 3mm punch biopsy is taken of the vaccine site. This is taken for laboratory analysis for immunohistochemical staining.
Other: Sterile water placement — 100mcg of sterile water will be administered intradermally on the back and serves as a negative control for the laboratory analysis. This will be injected intradermally on the back at 6 months post active immunization.

SUMMARY:
RATIONALE: Studying the immune response to a vaccine made from HER2/neu protein may help doctors plan better treatment for patients with breast cancer that overexpresses HER2.

PURPOSE: This clinical trial is studying the immune response in patients who have undergone vaccine therapy for stage III or stage IV breast cancer that overexpresses HER2.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether immunologic memory to the HER-2/neu (HER2) intracellular domain (ICD) protein has been generated by active immunization with a HER2 ICD plasmid-based vaccine by assessing the delayed-type hypersensitivity response to HER2 ICD peptides 6 months after vaccination in patients with HER2-overexpressing stage III or IV breast cancer.

Secondary

* Characterize the memory T-cell population and quantitate memory precursor frequency at 3, 6, and 12 months after active immunization using intracellular cytokine staining.

OUTLINE: This is an open-label study.

Patients receive HER2 intracellular domain (ICD) protein mixture intradermally and sterile water injected intradermally (as a negative control) at 6 months post-vaccination with pNGVL3-hICD vaccine. Vital signs and injection site will be monitored prior to skin test and at 60 minutes post-test. Patients return 48-72 hours after skin test for delayed-type hypersensitivity (DTH) measurements. The injection site is biopsied and examined by immunohistochemistry for infiltrating T-cell and antigen-presenting cell populations.

Blood is drawn at 3, 6, and 12 months post-vaccination for assessment of immune memory response. Blood draws are coordinated with parent study. Blood samples are examined by flow cytometry for the presence of memory markers including L-selectin, CD45 isoforms, cytokines, and CCR7.

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage III/IV breast cancer

  * Completed chemotherapy
  * Receiving trastuzumab (Herceptin®) monotherapy
* Successful completion of HER-2/neu (HER2) intracellular domain (ICD) plasmid-based vaccine trial (Protocol 01-9773-D06: "A Phase I Safety and Efficacy Trial of a DNA Plasmid Based Vaccine Encoding the HER-2/neu Intracellular Domain In Subjects With HER-2/neu-Overexpressing Tumors") within the past 3 months
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female (male patients are not excluded)
* Menopausal status not specified
* Zubrod performance status 0
* Unable to bear children (female patients)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No cytoreductive chemotherapy within the past 30 days
* No cytotoxic treatment and/or systemic corticosteroids within the past month
* Concurrent local radiotherapy or hormonal therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Immunologic memory response to HER-2/neu (HER2) intracellular domain protein | 6 months after active immunization

SECONDARY OUTCOMES:
Characterization of memory T-cell population by intracellular cytokine staining | 3, 6, and 12 months after active immunization
Quantitate memory precursor frequency by intracellular cytokine staining | 3, 6, and 12 months after active immunization

CONTACTS AND LOCATIONS:
Overall Officials: Lupe G. Salazar, MD, Principal Investigator — Tumor Vaccine Group at the University of Washington
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Tumor Vaccine Group at the University of Washington, Seattle, Washington